CLINICAL TRIAL: NCT05167045
Title: A Pilot Study for the Brain Health Support Program (BHSP) Intervention of the Canadian Therapeutic Platform Trial for Multidomain Interventions to Prevent Dementia
Brief Title: A Pilot Study for the Brain Health Support Program
Acronym: CTU BHSP-P
Status: Completed | Type: Observational
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Howard Chertkow, Scientific Director, Canadian Consortium on Neurodegeneration in Aging, Baycrest
Other Study IDs: CTU BHSP-P
Record Dates: First submitted 2021-11-01; First posted 2021-12-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Mild Cognitive Impairment; Subjective Cognitive Impairment; Pre-dementia; Dementia Prevention
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Dementia
  Interventions: Behavioral: Brain Health PRO

INTERVENTIONS:
Behavioral: Brain Health PRO — The BHSP is an educational program designed to teach about dementia. It aims to provide best available evidence for lifestyle changes that can help lower dementia risk, and to provide specific recommendations for positive lifestyle changes (e.g., physical exercises to try at home, healthy recipes). The program was developed as a collaborative effort by Canadian investigators who have expertise in the different areas of dementia prevention, along with input from older-adult citizen advisors.
  Other Names: Brain Health Support Program

SUMMARY:
Prior studies have shown that programs that focus on promoting brain health and managing lifestyle risks (such as poor diet, obesity, physical inactivity, sleep issues, loneliness) may help in preventing or lowering the risk of dementia. To address this, investigators have developed the CAN-THUMBS UP program to conduct studies that target lifestyle risk and focus on dementia prevention. An online Brain Health Support Program (BHSP) has been developed. The BHSP is an educational program designed to teach about dementia. Before the full BHSP is offered to a large group, we are conducting an initial pilot study to help assess the usability of the program.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for No Dementia and one of the following (according to CCNA criteria):

Cognitively Intact (CI) Cognitively Intact plus Subjective Cognitive Impairment (CI + SCI) Mild Cognitive Impairment (MCI)

• AND Classified as being at increased risk of dementia based on at least one of the following: First-degree family history of dementia

Self-Reported or documented current and/or history at midlife (45-60) on any of the following risk factors:

* Hypertension (documented Systolic Blood Pressure > 140 mm Hg; OR physician diagnosis of hypertension; OR treatment for hypertension; OR other approaches to treatment (e.g. diet, exercise))
* Hypercholesterolemia (documented total cholesterol > 6.5 mmol/L; OR physician diagnosis of hypercholesterolemia; OR treatment for hypercholesterolemia; OR other approaches to treatment (e.g. diet, exercise))
* Body Mass Index > 30 kg/m2 (derived from NIH Metric BMI Calculator)
* Physical Inactivity (active is defined as engaging in a minimum of 20- 30 min of physical activity causing sweating and breathlessness, at least 2 times a week)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit it's cohort from various locations around Canada.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Functionality of the BHSP | Nov 2021-Mar 2022
  Functionality of the web-based components of the BHSP measured in the pilot and qualitative focus group(s) questions
User acceptance of the BHSP | Nov 2021-Mar 2022
  User adherence and engagement using the online program during the pilot including dates and times of use, duration of use and completion of program assessments
Usability of the BHSP | Nov 2021-Mar 2022
  User satisfaction and evaluation of usability and acceptability of BHSP measured during the pilot and focus group(s)
To assess participant satisfaction with the organization, presentation and personalization of the BHSP content | Nov 2021-Mar 2022
  Qualitative evaluation of participant responses during the focus group discussion
To evaluate the feasibility of remote data collection | Nov 2021-Mar 2022
  User data, feedback and adherence to remote measures, such as: Screening evaluation by tele/video-conference, Neuropsychological Test Battery, Burst cognitive testing with the MyCogHealth app, online version of the Cogstate Brief Battery, Assessments of lifestyle risk factors (sleep, diet, mood, cognition, physical activity, vascular health, social and psychological health, vision and hearing), Actigraphy and EEG wearables as measures of total daily physical activity and sleep fragmentation, and Saliva sample collection for genomics testing (Polygenic Hazard Score)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of New Brunswick, Fredericton, New Brunswick
  - Baycrest, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Philip G, Fiocco AJ, Belleville S, Chertkow H, Feldman HH, Montero-Odasso M, Nygaard HB, Savundranayagam MY; Canadian Consortium on Neurodegeneration in Aging (CCNA), CAN-THUMBS UP Study Group. Exploring the usability and perceived benefits of Brain Health PRO: An online educational program for healthy brain aging. Digit Health. 2025 Nov 19;11:20552076251395585. doi: 10.1177/20552076251395585. eCollection 2025 Jan-Dec. PMID 41278371
- [Result] Belleville S, Anderson ND, Bherer L, Camicioli R, Carrier J, Chan S, Cuesta M, Dang-Vu TT, Dwosh E, Fiocco AJ, Ferland G, Gilbert B, Harris E, Itzhak I, Jarrett P, Kadri MA, Laurin D, Liu-Ambrose T, McGibbon CA, Middleton L, Miller L, Nygaard HB, Montero-Odasso M, Murphy K, Phillips N, Pichora-Fuller MK, Robillard JM, Smith EE, Speechley M, Trigui A, Wittich W, Chertkow H, Feldman HH; CTU expert group for the Canadian Consortium on Neurodegeneration in Aging (CCNA), CAN-THUMBS UP Study Group. Brain health PRO/Sante cerveau PRO: The development of a web-based program for dementia literacy and risk factor reduction. J Prev Alzheimers Dis. 2025 Jun;12(6):100134. doi: 10.1016/j.tjpad.2025.100134. Epub 2025 Mar 15. PMID 40090784